CLINICAL TRIAL: NCT00469794
Title: The Long Term Significance of Exercise Induced Ventricular Arrhythmias in Trained Athletes
Brief Title: The Significance of Arrhythmias in Athletes
Acronym: Athlete
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Institute of Physical Education and Sports Sciences (Other)
Other Study IDs: 50/06
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Sudden Death
Keywords: arrhythmias; Athletes; exercise
MeSH Terms: conditions — Death, Sudden; Arrhythmias, Cardiac; Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: stress test

SUMMARY:
Athletes with complex ventricular arrhythmias are potentially at risk of sudden death. The aim of the study is to investigate the relevance of ventricular tachyarrhythmias induced by an exercise test in a retrospectively evaluated athletic population.

DETAILED DESCRIPTION:
Athletes with complex ventricular arrhythmias are potentially at risk of sudden death. The risk is increased when the athletes are engaged in competitive activities.

Ventricular premature beats (VPB's) are a common finding in the athletic heart. In the majority of cases these arrhythmias are part of the "athlete's heart syndrome" and do not increase the risk of sudden death in the athletes with an apparently normal heart. The data available in the literature deal with ventricular arrhythmias assessed only by 24-h ambulatory electrocardiograms.

To date, there are no guidelines concerning athletes who develop ventricular arrhythmias during a stress test. It is unclear whether they should be allowed to continue with their competitive activity or they should be denied to do so. A study looking at the long term follow-up of these athletes will help us determine whether the development of ventricular arrhythmia during a stress test imposes any risk on the athletes.

ELIGIBILITY:
Inclusion Criteria:

* Competitive athletes less than 35 YO
* Competitive athletes with ventricular arrhythmias on baseline or recovery in a stress test
* Competitive athletes with ventricular arrhythmia during exercise

Exclusion Criteria:

* Athletes who don't meet the exclusion criteria.

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-05; Study Completion 2008-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Therese Fuchs, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Wingate Institute, Netanya, Israel